CLINICAL TRIAL: NCT03556436
Title: An Open-label, Single-dose Phase 1 Clinical Trial to Evaluate the Safety and Effects of Ethnicity and Food on Pharmacokinetics of YH25448 in Healthy Korean and Caucasian Volunteers
Brief Title: Clinical Trial to Evaluate the Safety and Effects of Ethnicity and Food on Pharmacokinetics of YH25448
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YH25448-101
Record Dates: First submitted 2018-06-01; First posted 2018-06-14 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: YH25448; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): YH25448 240mg single dose in korean
  Interventions: Drug: YH25448 240mg
- Group 2 (Experimental): YH25448 240mg single dose in caucasian
  Interventions: Drug: YH25448 240mg

INTERVENTIONS:
Drug: YH25448 240mg — period 1: A single oral dose of YH25448 240 mg an overnight fast period 2: A single oral dose of YH25448 240 mg after a high-fat breakfast
  Other Names: YH25448

SUMMARY:
Clinical trial is to evaluate the effect of ethnicity and food on the pharmacokinetics (how a drug is absorbed, metabolized, distributed and excreted; plasma drug concentration will be measured in this clinical trial) of YH25448, which Yuhan Corporation plans to develop as a therapeutic agent for Non-Small Cell Lung Cancer.

DETAILED DESCRIPTION:
This clinical trial will be conducted in healthy Korean and Caucasian volunteers at Seoul National University Hospital (SNUH) Clinical Trial Center.

It is expected to take approximately 39 days from the first dosing of Investigational Product until the final follow-up visit. It will be hospitalized twice for 9 nights and 10 days with 21 days of interval, and one visit will be needed for safety evaluation between 14-17 days from the last dosing of the Investigational Product.

ELIGIBILITY:
Inclusion Criteria:

1. Informed of the investigational nature of this study and voluntarily agree to participate in this study.
2. Subjects with BMI range of ≥18.5 kg/m2 and < 30.0 kg/m2 and weighing ≥ 50 kg
3. Subjects without congenital or chronic diseases within the last 3 years and without pathologic symptoms as determined by medical diagnosis
4. Healthy Korean and Caucasian males who aged ≥ 19 and ≤ 55 years at the time of consent

Exclusion Criteria:

1. Clinically significant chronic infection (e.g. AIDS) or clinically significant medical or psychiatric illness
2. Hypotension (SBP ≤ 90 mmHg or DBP ≤ 50 mmHg) or hypertension (SBP ≥ 150 mmHg or DBP ≥ 100 mmHg)
3. A marked baseline prolongation of QTc greater than 450 msec by Bazett's formula
4. Within 14 days prior to the first administration of investigational product, use of prescription drugs or herbal medication, or within 7 days use of any over-the-counter medications

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
AUClast of YH25448 | 0-192 hrs
  Area under the plasma concentration-time curve from zero to the time of the last quantitative concentration (AUC) of YH25448
Cmax of YH25448 | 0-192 hrs
  Area under the plasma concentration-time curve from zero to the time of Maximum plasma concentration (Cmax) of YH25448

SECONDARY OUTCOMES:
AUCinf of YH25448 | 0-192 hrs
  Area under the plasma concentration time curve from zero to infinity (AUC) of YH25448
Tmax of YH25448 | 0-192 hrs
  Time to reach Cmax of YH25448
t1/2 of YH25448 | 0-192 hrs
  Terminal half life (t1/2) of YH25448
CL/F of YH25448 | 0-192 hrs
  The apparent plasma clearance (CL/F) of YH25448
Vd/F of YH25448 | 0-192 hrs
  Apparent Volume of distribution of YH25448

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital Clinical Trial Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No